CLINICAL TRIAL: NCT00378859
Title: The Effect of Milk and Meat on IGFs in Prepubertal Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KF 01-097/00; D-110
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-09

CONDITIONS: Growth Disorders; Metabolic Syndrome
Keywords: Children; Milk; Meat; Animal Protein; Growth Factors; IGF-I; IGFBP-3; Insulin
MeSH Terms: conditions — Growth Disorders; Metabolic Syndrome; Insulin Resistance

INTERVENTIONS:
Behavioral: Skim milk
Behavioral: Lean meat

SUMMARY:
The objective of the study is to examine whether a 7-day high protein intake from either milk or meat in healthy, prepubertal children can increase fasting levels of serum IGF-I, IGFBP-3 and IGF-I/IGFBP-3 as well as insulin, glucose and HOMA insulin reststance, HOMA beta cell function and amino acids.

DETAILED DESCRIPTION:
The objective of the study is to examine whether a high protein intake (PI) from either milk or meat, at a level often seen in late infancy, in healthy, prepubertal children can increase fasting levels of serum IGF-I, IGFBP-3 and IGF-I/IGFBP-3 as well as insulin, glucose and HOMA insulin reststance, HOMA beta cell function and amino acids.

IGF-I levels are positively associated with growth velocity in children and some studies suggest that a high animal PI can stimulate growth. During protein deprivation IGF-I decrease, but it is unknown whether a high PI can increase s-IGF-I in well-nourished children.

Insulin is also a growth factor, and studies have found that postprandially, milk possess some insulinotrophic effect not related to its carbohydrate content. However, the effect on fasting insulin in children is unknown.

Design: Twenty-four 8-y-old boys are asked to take either 1.5 l of skimmed milk (n=12) or the same amount of protein as 250 g low fat meat (n=12) daily for seven days. The remaining diet they can choose freely. At baseline and after seven days, anthropometrical variables are measured, diet is registered (3-d weighed records), and the blood analytes are determined after fast.

ELIGIBILITY:
Inclusion Criteria:

* habital milk intake more than 500 mL/d
* willing to increase intake of milk or meat considerably for one week

Exclusion Criteria:

* chronic illnesses
* children who suffer from any condition likely to affect their protein metabolism or growth

Ages: 8 Years to 8 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24
Dates: Start 2000-11; Study Completion 2001-03

PRIMARY OUTCOMES:
IGF-I
IGFBP-3
Insulin
Glucose
Aminogram

SECONDARY OUTCOMES:
Blood Pressure
Kidney Size
Urea Nitrogen
Adiponectin
Leptin
Ghrelin
Osteocalcin
BAP
CTX

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Dr Med Sci, Study Chair — Institute of Human Nutrition, Rolighedsvej 30, DK-1958 Frederiksberg C, Denmark
Locations (1):
- Institute of Human Nutrition, Rolighedsvej 30, Frederiksberg C, Denmark